CLINICAL TRIAL: NCT05210348
Title: Clinical Evaluation Study of Urine hrHPV Detection for the Diagnosis of Presence of Cervical HPV and Correlation of Cervical Lesions
Brief Title: Clinical Evaluation of Detection of High Risk HPV in Urine
Acronym: Urine-hrHPV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Hangzhou Mingze Medical Research Co., Ltd. (Unknown); Beijing Tsingke Biological Technology Co., Ltd. Hangzhou Branch (Unknown); Hangzhou Newhorizon Health Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Wang Jianliu, Chief physician, Peking University People's Hospital
Other Study IDs: Urine-hrHPV 2021
Record Dates: First submitted 2022-01-07; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-12

CONDITIONS: Human Papillomavirus Infection; Cervical Cancer; Human Papilloma Virus; Negative for Intraepithelial Lesion or Malignancy; Atypical Squamous Cells of Undetermined Significance; Cervical Squamous Intraepithelial Lesion; Atypical Squamous Cells, Cannot Rule Out High-grade Squamous Intraepithelial Lesion; Low-grade Squamous Intraepithelial Lesion; High-Grade Squamous Intraepithelial Lesions; Cervical Intraepithelial Neoplasia Grade I; Cervical Intraepithelial Neoplasia Grade II; Cervical Intraepithelial Neoplasia, Grade III; Atypical Glandular Cells; Atypical Glandular Cells Not Otherwise Specified; Atypical Glandular Cells, Favor Neoplastic; Cervical Squamous Cell Carcinoma; Adenocarcinoma in Situ; Cervical Adenocarcinoma
Keywords: Urine testing for high-risk HPV; Human papilloma virus; Cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Neoplasms; Atypical Squamous Cells of the Cervix; Squamous Intraepithelial Lesions; Uterine Cervical Dysplasia; Adenocarcinoma in Situ

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HPV positive group
- HPV negative group
- Disease group (clinical diagnosis positive): CIN2 and above disease cases, including HSIL or (CIN2, CIN2-3, CIN3) cervical cancer.
- Control group (clinical diagnosis is negative): includes other benign lesions such as inflammation, polyps, and HPV-negative cases without pathological diagnosis and no abnormalities in TCT.

SUMMARY:
Cervical cancer is one of the most common tumors in women, which seriously threatens women's life quality and safety. Human papilloma virus (HPV) infection is the most common cause of cervical cancer. Traditional HPV testing is based on the cells sample shed from the cervix. Recent studies have shown that urine HPV detection can be used as a new HPV detection method. This study intends to include patients undergoing TCT /HPV test/colposcopy in the department of gynecological diseases of the hospital, and collect urine samples and cervical swab samples. Sanger sequencing and cervical swab HPV test results were compared to evaluate the accuracy and clinical validity of urine HPV test combined with clinical diagnosis results of cases.

DETAILED DESCRIPTION:
The urine high-risk HPV detection reagent (PCR-fluorescent probe method) developed by Hangzhou Newhorizon Health Technology Co., Ltd. can qualitatively detect 14 high-risk HPV DNA in human urine samples, including HPV16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68, and can detect HPV 16 and 18.

This test adopts the comparative clinical research method, by collecting urine samples and cervical swab samples from the same subject for HPV nucleic acid detection. Among them, urine samples were tested for high-risk HPV nucleic acid testing and Sanger sequencing, and cervical swab samples were tested with HPV testing kits for cervical swabs that have been on the market. Combined with the clinical diagnosis results of the cases, the performance of the urine HPV detection technology is compared and evaluated.

For patients undergoing TCT testing/HPV testing/colposcopy in the gynecological clinic or colposcopy clinic of the hospital, the subjects will be screened through the admission criteria and signed an informed consent; the examiner is required to collect cervical swab samples and, at the same time, issue urine collection When the tube is given to the subject, the subject must collect urine samples by themselves according to the sampling instructions or under the guidance of medical personnel; the patient samples will be tested by Hangzhou Newhorizon Health Technology Co., Ltd.; the clinical examination report will be collected as the case materials of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20-65 years old;
2. Have a history of sexual life;
3. The patients were voluntarily enrolled in the group and signed an informed consent form.

Exclusion Criteria:

1. History of cervical conization, pelvic radiation and hysterectomy, acute inflammation of the reproductive tract, severe system disease or other malignant tumors;
2. Pregnant and lactating women;
3. The patient's compliance is poor or the researcher thinks it is not suitable for this study.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing TCT/HPV/colposcopy in the gynecological clinic or colposcopy clinic of the hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Verification of accuracy | 2022/5
  Consistency analysis of urine HPV test and Sanger sequencing results/cervical swab HPV test results The main evaluation indicators are the total test positive coincidence rate, total test negative coincidence rate, total coincidence rate, 16/18/other 12 types of positive and negative coincidence rates, kappa value and 95% confidence interval.

SECONDARY OUTCOMES:
Clinical validity verification | 2022/5
  Using the clinical diagnosis result (colposcopy or pathology report) of the case as the gold standard, evaluate the sensitivity, specificity and the corresponding 95% confidence interval, etc. of the HPV detection of urine samples and cervical swab samples for cervical intraepithelial neoplasia grade II and above (≥CIN2)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanjing First Hospital, Nanjing, Jiangsu

REFERENCES:
- [Background] Arbyn M, Castellsague X, de Sanjose S, Bruni L, Saraiya M, Bray F, Ferlay J. Worldwide burden of cervical cancer in 2008. Ann Oncol. 2011 Dec;22(12):2675-2686. doi: 10.1093/annonc/mdr015. Epub 2011 Apr 6. PMID 21471563
- [Background] Saxena U, Sauvaget C, Sankaranarayanan R. Evidence-based screening, early diagnosis and treatment strategy of cervical cancer for national policy in low- resource countries: example of India. Asian Pac J Cancer Prev. 2012;13(4):1699-703. doi: 10.7314/apjcp.2012.13.4.1699. PMID 22799391
- [Background] Bosch FX, Lorincz A, Munoz N, Meijer CJ, Shah KV. The causal relation between human papillomavirus and cervical cancer. J Clin Pathol. 2002 Apr;55(4):244-65. doi: 10.1136/jcp.55.4.244. PMID 11919208
- [Background] Walboomers JM, Jacobs MV, Manos MM, Bosch FX, Kummer JA, Shah KV, Snijders PJ, Peto J, Meijer CJ, Munoz N. Human papillomavirus is a necessary cause of invasive cervical cancer worldwide. J Pathol. 1999 Sep;189(1):12-9. doi: 10.1002/(SICI)1096-9896(199909)189:13.0.CO;2-F. PMID 10451482
- [Background] Munoz N, Bosch FX, de Sanjose S, Herrero R, Castellsague X, Shah KV, Snijders PJ, Meijer CJ; International Agency for Research on Cancer Multicenter Cervical Cancer Study Group. Epidemiologic classification of human papillomavirus types associated with cervical cancer. N Engl J Med. 2003 Feb 6;348(6):518-27. doi: 10.1056/NEJMoa021641. PMID 12571259
- [Background] Khan MJ, Castle PE, Lorincz AT, Wacholder S, Sherman M, Scott DR, Rush BB, Glass AG, Schiffman M. The elevated 10-year risk of cervical precancer and cancer in women with human papillomavirus (HPV) type 16 or 18 and the possible utility of type-specific HPV testing in clinical practice. J Natl Cancer Inst. 2005 Jul 20;97(14):1072-9. doi: 10.1093/jnci/dji187. PMID 16030305
- [Background] zur Hausen H. Papillomaviruses in the causation of human cancers - a brief historical account. Virology. 2009 Feb 20;384(2):260-5. doi: 10.1016/j.virol.2008.11.046. Epub 2009 Jan 8. PMID 19135222
- [Background] Pinto AP, Crum CP. Natural history of cervical neoplasia: defining progression and its consequence. Clin Obstet Gynecol. 2000 Jun;43(2):352-62. doi: 10.1097/00003081-200006000-00015. No abstract available. PMID 10863633
- [Background] Bernal S, Palomares JC, Artura A, Parra M, Cabezas JL, Robles A, Martin Mazuelos E. Comparison of urine and cervical samples for detecting human papillomavirus (HPV) with the Cobas 4800 HPV test. J Clin Virol. 2014 Dec;61(4):548-52. doi: 10.1016/j.jcv.2014.10.001. Epub 2014 Oct 12. PMID 25453566
- [Background] Hagihara M, Yamagishi Y, Izumi K, Miyazaki N, Suzuki T, Kato H, Nishiyama N, Koizumi Y, Suematsu H, Mikamo H. Comparison of initial stream urine samples and cervical samples for detection of human papillomavirus. J Infect Chemother. 2016 Aug;22(8):559-62. doi: 10.1016/j.jiac.2016.05.009. Epub 2016 Jun 21. PMID 27342077
- [Background] Pathak N, Dodds J, Zamora J, Khan K. Accuracy of urinary human papillomavirus testing for presence of cervical HPV: systematic review and meta-analysis. BMJ. 2014 Sep 16;349:g5264. doi: 10.1136/bmj.g5264. PMID 25232064
- [Background] Combita AL, Gheit T, Gonzalez P, Puerto D, Murillo RH, Montoya L, Vorsters A, Van Keer S, Van Damme P, Tommasino M, Hernandez-Suarez G, Sanchez L, Herrero R, Wiesner C. Comparison between Urine and Cervical Samples for HPV DNA Detection and Typing in Young Women in Colombia. Cancer Prev Res (Phila). 2016 Sep;9(9):766-71. doi: 10.1158/1940-6207.CAPR-16-0038. Epub 2016 Jul 14. PMID 27417431
- See also: Related Info — http://rs.yiigle.com/CN119273201601/866671.htm